CLINICAL TRIAL: NCT02459639
Title: Existential Genomics (ExiGence): Effects of Multimodal Rehabilitation and Integrative Care on Pain, Quality of Life, and Genomic Stability in Patients With Chronic Pain
Brief Title: Existential Genomics: Effects of Multimodal Rehabilitation and Integrative Care on Patients With Chronic Pain
Acronym: ExiGence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Integrative Care Science Center (Other)
Collaborators: University Hospital, Linkoeping (Other); Ekhagastiftelsen (Other)
Responsible Party: Principal Investigator, Torkel Falkenberg, Associate Professor, The Integrative Care Science Center
Other Study IDs: 2014-37
Record Dates: First submitted 2015-05-21; First posted 2015-06-02 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Pain
Keywords: Chronic Widespread Pain; Telomere length; Multimodal rehabilitation; Integrative care; Existential aspects
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Leucocyte cell extracts
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anthroposophic integrative care: Inclusion criteria are: Pain patients with a primary diagnosis corresponding to ICD-10 M79, or long-term pain for a period of over 3 months in neck/shoulders and/or low back, or generalised pain, fluency in Swedish and allowing for co-morbidity/ multiple secondary diagnoses.
  The exclusion criteria are: psychotic illness, schizophrenia, bipolar disorder, substance dependency problems, and cancer.
  Interventions: Other: Anthroposophic integrative care rehabilitation program
- Multimodal pain rehabilitation: Inclusion criteria are: Pain patients with a primary diagnosis corresponding to ICD-10 M79, or long-term pain for a period of over 3 months in neck/shoulders and/or low back, or generalised pain, fluency in Swedish and allowing for co-morbidity/ multiple secondary diagnoses.
  The exclusion criteria are: psychotic illness, schizophrenia, bipolar disorder, substance dependency problems, and cancer.
  Interventions: Other: Conventional multi-modal care rehabilitation

INTERVENTIONS:
Other: Anthroposophic integrative care rehabilitation program — The programme for chronic pain at AIC consists of two phases:
  1. A three-week in-patient period. During the first three-week in-patient stay, patients meet regularly with a multi-professional team. Usually, each patient receives two of the following therapies 2-4 times per week: art therapy, massage, physiotherapy, eurhythmy and baths. Nursing care is provided twice daily. Moreover, patients are offered to participate in group activities.
  2. Two-three day inpatient follow-up and treatment period closure. The second phase of the treatment programme consists of a 2-3 day inpatient stay, 6 months after closure. During this time, physician, nurse and therapist appointments are made according to individual needs. The patients who have been engaged in group activities are gathered in groups.
  Groups: Anthroposophic integrative care
Other: Conventional multi-modal care rehabilitation — The standard approach at Linköping University Hospital admits patients for bio-psycho-social assessment, pharmacological treatment and multimodal rehabilitation (main components: education, intense physical exercise, cognitive behavioural therapy and workplace interventions) for a 6 week intensive phase period (75%) followed by 4 weeks (25%). Here a number of professional disciplines collaborate and form a team of professionals focused on individual patient needs The multimodal rehabilitation outpatient program delivered by this team has the following aims: 1) reduce pain and psychological burden, 2) improve work capacity and decrease sick-leave and 3) increase perceived health and quality of life. These general aims are combined with the aims of the patient in a plan of rehabilitation.
  Groups: Multimodal pain rehabilitation

SUMMARY:
Using a comprehensive prospective clinical study design, the investigators intend to compare changes in health-related markers in patients with chronic widespread pain (CWP), undergoing one of two intervention "packages" of multimodal health care, namely anthroposophical integrative care (AIC) or standard care (SC), respectively. AIC combines evidence-based conventional care with complementary/alternative (CAM) treatments. As markers, the investigators will use indicators of drug utilization and sick leave, as well as constructs mirroring possible changes in psychological and existential factors and genomic stability (such as telomere length and telomerase levels).

DETAILED DESCRIPTION:
The purpose of this comprehensive prospective clinical study is to compare and contrast two different but well-established multimodal chronic widespread pain rehabilitation programmes, i.e. one at a conventional county council hospital (CC) and one involving integrative care at a private non-profit hospital (IC), in terms of changes in health-related outcomes, ranging from DNA stability to health economy, in patients with chronic pain. Notably, for the first time, differences can be seen and correlations made between CC and IC outcomes with relevance for clinical care development and implementation of multimodal interventions for people with chronic pain.

The overall aim of the present prospective clinical trial is to achieve a better understanding of the possible effects of, and useful measure for evaluating, two different multimodal treatment interventions for pain.

More specifically, the aims of this trial are to explore two different, but well-established multimodal pain rehabilitation programmes. The investigators will specifically investigate 1. If chronic pain impacts on patients' telomerase activity and telomere length over time; 2. If multimodal rehabilitation can be linked to positive changes in telomerase activity and telomere length after rehabilitation, and if these changes can be correlated to: Clinical diagnosis, pain characteristics (e.g. intensity, duration, frequency and spread of pain), co-morbidities (e.g. anxiety, depression and catastrophizing), time lost from work/sick-leave and self-rated health and stress, and; 3. If and how the two programmes and their treatment components differ in outcomes over time.

The project outcomes will be of great relevance for clinical rehabilitation development and the implementation of multimodal interventions for people with chronic pain. Given that the most significant demographic and clinical factors associated with pain help-seeking are increasing age, female gender, pain severity and disability, we will also address such issues including gender differences when relevant.

Specific work packages (WP): WP1 - Genomics (telomerase activity and telomere length); WP2 - Patient-reported outcomes ("existential" validated questionnaires regarding depression, anxiety, stress, quality of life, pain, mindfulness, spirituality/religiosity); WP3 - Health care experiences (interviews); WP4 - Registry data (drugs, health care, sick leave, return-to-work, morbidity, mortality); WP5 - The design of treatment programs; WP6 - Standardized and exploratory statistical analyses of differences and correlations between the collected data and the conventional and integrated care programs. WP7 - Implementation of the results problematized through the participation of representatives of the patient and care provider organizations.

ELIGIBILITY:
Inclusion Criteria:

* Pain patients with a primary diagnosis corresponding to ICD-10 M79, or long-term pain for a period of over 3 months in neck/shoulders and/or low back, or generalised pain,
* fluency in Swedish and
* allowing for co-morbidity/ multiple secondary diagnoses.

Exclusion Criteria:

* Psychotic illness,
* schizophrenia,
* bipolar disorder,
* substance dependency problems, and
* cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 pain patients will be recruited into the study. They will be invited to participate in the study upon admission to Integrative Care pain rehabilitation at the Vidar Clinic (n=50) or the Pain Clinic, University Hospital, Linköping (n=50).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Telomere length from blood sample leucocyte cells | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  telomere length from blood sample leucocyte cells
Telomerase activity from blood sample leucocyte cells | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  telomerase activity from blood sample leucocyte cells

SECONDARY OUTCOMES:
Hb - hemoglobin status | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  blood hemoglobin status
Cholesterol: Blood cholesterol levels | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  Blood cholesterol levels
C-Reactive Protein levels in blood sample | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  C-Reactive Protein
Trigyceride levels in blood sample | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  Triglyceride levels in blood sample
Glucose levels in blood sample | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  Glucose levels in blood sample
LDL-cholesterol levels in blood sample | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  LDL-cholesterol levels in blood sample
HDL-cholesterol levels in blood sample | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  HDL-cholesterol levels in blood sample
Blood pressure | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  Resting systolic and diastolic blood pressure
Body Mass Index | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  Body Mass Index calculated from weight and length
Chronic Pain Acceptance Questionnaire - 8: measuring acceptance of chronic pain | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  8 question questionnaire assessing self-rated chronic pain acceptance, numerical total score
Five Facet Mindfulness Questionnaire: measuring level of mindfulness | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  29 questionnaire assessing self-rated mindfulness, numerical composite score
Hospital Anxiety and Depression scale: measuring level of anxiety and depression | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  self-rating scale for assessing anxiety and depression levels, numeric total score
EuroQol 5 Dimensions: measuring health-related quality of life | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  salf-rating scale for health-related quality of life, numeric total score
Indicator Questions of Physical Activity: measuring level of physical activity | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  Self-rated assessment of physical activity, three questions, numeric total score
sociodemographic questionnaire | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  baseline and follow-up sociodemographic questionnaire from NRS (Nationalle Registret över Smärtrehabilitering), numeric descriptive data
WHO Quality of Life - Spiritual, Religious and Personal Beliefs | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  a medium- length 37 question version of a self-rating scale for quality of life, spiritual, religious and personal beliefs, numeric total score
Use of prescription drugs | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  register-based data on use of prescription drugs, dose and frequency
Sick-leave data | baseline, up to 6 weeks, 6 month-, and 1 year follow-up
  register-based data on sick-leave, extent and time period
patient records | up to 6 weeks and 1 year follow-up
  treatment records on the treatment components obtained by patient, amount and frequency

CONTACTS AND LOCATIONS:
Overall Officials: Torkel Falkenberg, Ass. Prof, Principal Investigator — Integrative Care Science Center

REFERENCES:
- [Derived] Ronne-Petersen L, Niemi M, Walach H, Lavebratt C, Yang LL, Gerdle B, Ghafouri B, Falkenberg T. Exploring emotional well-being, spiritual, religious and personal beliefs and telomere length in chronic pain patients-A pilot study with cross-sectional design. PLoS One. 2024 Sep 4;19(9):e0308924. doi: 10.1371/journal.pone.0308924. eCollection 2024. PMID 39231146